CLINICAL TRIAL: NCT01518296
Title: Rating the Degree of Pelvic Organs Prolapse in Women According to the POPQ Method Before and After Emptying the Urinary Bladder
Brief Title: Rating Pelvic Organs Prolapse in Women According to the POPQ Method Before and After Emptying the Urinary Bladder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Eran Segev, Resident in Ob/Gyn department, Camel Medical Center, Carmel Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CMC-11-0071-CTIL
Record Dates: First submitted 2012-01-22; First posted 2012-01-25 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Patients With Pelvic Organs Prolapse
Keywords: Pelvic Organ Prolapse Quantification (POPQ); POPQ; Urodynamic test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients referred to urodynamic test (Experimental): Patients that are referred to urogynecology and the pelvic reconstruction unit undergoes a physical gynecological examination and a urodynamic test, During which the degree of pelvic organs prolapse is evaluated with full and empty bladder.
  Interventions: Device: Medtronic-Dantec Urodynamic System

INTERVENTIONS:
Device: Medtronic-Dantec Urodynamic System — Urodynamic test is test performed in order to assess whether there is a urinary incontinence and underlying cause. During this test the woman is asked to empty her bladder and then two transducers are inserted, one into the bladder and the other into the rectum, then the bladder is filled with physiological solution and the patient is asked to urinate. During bladder emptying urinary flow velocity is measured and the pressures in the abdomen and bladder are recorded for later evaluation

SUMMARY:
Pelvic organ prolapse is a common disorder that affects 3-9% of adult women. Treatment of this disorder varies and includes conservative and interventional treatment.

Pelvic organs prolapse grading has an important roll in determining the appropriate treatment. Developments in this field has led to the development of an agreed method to rate the degree of pelvic organs prolapse (POPQ).

The roll of Urodynamic test is to assess whether there is urinary incontinence and underlying cause.

In Richard C. et al publication, that presented the Pelvic Organ Prolapse Quantification (POPQ) method for the first time, there was no reference to the urinary bladder state (full or empty) during the examination, hence the investigators are asking to conduct a prospective study in order to evaluate the degree of pelvic organs prolapse according to POPQ method during urodynamic examination, with a full and empty urinary bladder.

DETAILED DESCRIPTION:
Pelvic organ prolapse is a common disorder that affects 3-9% of adult women. Treatment of this disorder varies and includes behavioral therapy, pelvic floor muscles rehabilitation exercises, medication therapy, devices that are tailored to the patient in order to improve pelvic organ support and various surgical procedures. Developments in this field and the need to tailor the appropriate treatment to the type and degree of pelvic organ prolapse resulted in the development of an agreed method to rate the degree of pelvic organs prolapse.

Pelvic organs prolapse grading has an important roll in determining the appropriate treatment. A big proportion of women who suffer from pelvic organ prolapse suffer from urinary system disorders as well, such as difficulty in urinating, urinary incontinence, and urgency and frequency.

At the pelvic floor reconstruction clinic, women who suffer from pelvic organs prolapse, undergo a preliminary workup that includes a medical questionnaire, physical examination to evaluate the degree of pelvic organ prolapse according to the Pelvic Organ Prolapse Quantification method (POPQ), and a urodynamic test.

The impression of differences in the degree of prolapse according to POPQ method, before and after urination, has led to the hypothesis that the degree of pelvic organs prolapse varies according to the degree of fullness of the bladder

Urodynamic test is a test performed during patient evaluation at the pelvic floor reconstruction clinic. During this test the woman is asked to empty her bladder and then two transducers are inserted, one into the bladder and the other into the rectum. During the test the bladder is filled with physiological solution and then the patient is asked to urinate. During bladder emptying urinary flow velocity is measured and the pressure in the abdomen and bladder recorded for later evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Women with pelvic organs prolapse
2. Women who can read and understand and sign consent form
3. Women between 20 and 90 years of age.

Exclusion Criteria:

1. Women who underwent vaginal gynecologic surgery in the past
2. women that underwent hysterectomy

Ages: 20 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Evaluating the degree of pelvic organs prolapse according to POPQ method, with filled and empty urinary bladder, during urodynamic test | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Eran Segev, MD, Principal Investigator — Carmel Medical Center
Locations (1):
- Carmel Medical Center, Haifa, Israel